CLINICAL TRIAL: NCT05683431
Title: Bipolar Remediation of Affective Impulsivity and Negative Symptomatology (BRAINS)
Brief Title: Using Neuroplasticity-Based Computerized Training to Improve Emotion Regulation in Bipolar Disorder (BRAINS)
Acronym: BRAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: The Ryan Licht Sang Bipolar Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17042901
Record Dates: First submitted 2018-04-23; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Bipolar Disorder; Bipolar I Disorder; Bipolar Affective Disorder; Bipolar Disorder I; Bipolar Depression
Keywords: Bipolar; Emotion; Cognitive Control; Affect; Impulsivity; Neuroimaging; Targeted Cognitive Training
MeSH Terms: conditions — Bipolar Disorder; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: This is a single-arm, 'open label' study to examine the feasibility and potential target engagement (i.e. potential benefit) of a behavioral smartphone-based cognitive training program for individuals with bipolar I disorder. Participants with bipolar disorder are assessed before and after the 20 session/4 week intervention. In addition, a comparison group of healthy adults (without bipolar disorder) are assessed at a single time-point as a means of identifying baseline deficits associated with bipolar disorder. Participants in the healthy comparison group do not complete the intervention. (Thus, Number of Intervention Arms = 1.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Control of Emotion (CCE) Training (Experimental): Mobile (iphone/ipad) "App" with game-like exercises designed to improve Cognitive Control of Emotion (CCE), i.e. the ability to control the influence of emotional information on behavior. Participants do 20 sessions (approximately 30min each), over 4 weeks.
  Interventions: Behavioral: Cognitive Control of Emotion (CCE) Training

INTERVENTIONS:
Behavioral: Cognitive Control of Emotion (CCE) Training — Training consists of game-like exercises using a software program developed in collaboration with PositScience Corporation (using BrainHQ platform ) - which has exercises targeting cognition and social cognition. The CCE training program incorporates characteristics that optimize learning-induced neuroplasticity - most importantly, exercises are short & rewarding, adapt to individual skill-level, and become increasingly difficult as performance improves. There are 5 CCE exercises that are organized in half-hour sessions and proceed in a predetermined sequence.
  Other Names: Cognitive Control of Emotion Training using a BrainHQ smartphone "App" developed by Posit Science

SUMMARY:
The goal of this study is to evaluate the feasibility and potential benefit of a behavioral intervention designed to improve emotion regulation in individuals with bipolar disorder. The intervention consists of game-like exercises that involve the 'Cognitive Control of Emotion (CCE) - i.e. the ability to control the influence of emotional information on behavior. Deficits in the cognitive control of emotion are a central feature of Bipolar Disorder that contributes to emotion dysregulation, maladaptive mood episodes, and, ultimately, the overall chronicity and severity of illness. Neuroimaging studies of bipolar patients demonstrate neural abnormalities in brain systems involved in cognitive control and emotion processing. Furthermore, these abnormalities predict mood and behavior problems associated with cognitive control of emotion, such as emotion lability, disinhibited behavior, and extreme mood states. The aim of this study is to determine feasibility and examine whether a computer-based program of progressively difficult cognitive control emotion exercises will improve cognitive control of emotion skills and, thereby, result in better emotion regulation and daily functioning in young adults with bipolar disorder. To test the intervention, a single group of young adults (18-30 years old) with Bipolar I Disorder will complete behavioral assessments before and after 20 hours (4 weeks) of CCE training. In order to identify baseline deficits associated with bipolar disorder, a comparison group of healthy young adults will complete behavioral assessments at a single time-point (without CCE training).

DETAILED DESCRIPTION:
Difficulty with emotion regulation is a central feature of Bipolar Disorder (BD) that is not only apparent during mood episodes but also persists in between episodes and contributes to the onset, chronicity, and severity illness. Successful emotion regulation requires the cognitive control of emotion (CCE) - i.e. the ability to control emotions and the influence of emotions on behavior. CCE is dependent on the coordinated activity of two neural systems: 1) the cognitive control network includes the lateral prefrontal cortex and superior parietal cortex and supports a range of skills (e.g. attention, inhibition, working memory) to control and manipulate information from multiple sensory domains; and 2) the emotion processing network, which includes the amygdala, insula, and ventral striatum, and supports the experience, expression, and perception of emotion. CCE consists of several processes in which the cognitive control network modulates neural response in emotion processing regions to control the impact of emotion on experience and behavior. Poor recruitment of frontoparietal control functions when processing negative emotional stimuli (measured with fMRI) prospectively predicts mood and behavioral problems after an interpersonal conflict in daily life (Hooker et al 2010). Together the data suggests that compromised CCE capacity makes a person more vulnerable to experiencing negative psychological consequences after a stressful event (e.g. Hooker et al 2010; Hooker et al 2013; Tully et al 2014).

Individuals with bipolar disorder have deficits on both behavioral and neural measures of CCE (Phillips and Swartz 2014). Typical CCE tasks require identifying a target stimulus (e.g. word, facial expression, etc.) while inhibiting irrelevant or conflicting emotional information. During such tasks, people with bipolar disorder have difficulty controlling the distracting influence of irrelevant emotional information. These behavioral deficits are associated with neural abnormalities in both cognitive control and emotion processing neural systems. These neural abnormalities are characterized, primarily, by abnormally low activity in the cognitive control network, particularly the lateral prefrontal cortex, and abnormally high activity in emotion processing regions, particularly the amygdala and ventral striatum. Bipolar disorder is also associated with abnormalities in structural elements of these neural systems, including abnormal gray matter volume and white matter tracks. Research suggests that deficits in CCE and related neural networks are an underlying cause of characteristic symptoms of bipolar disorder, including emotional lability, extreme mood states, and disinhibited behavior (reviewed in Phillips and Swartz 2014 and Wegbreit et al. 2014). These findings point to CCE as a clinically relevant and scientifically tractable treatment target for bipolar.

Study Design & Specific Aims The primary goal of this project is to investigate, in young adults with bipolar disorder, whether a computerized training program of CCE exercises improves CCE as measured with a range of assessment tasks that require flexible deployment of CCE skills. The long-term goal is to evaluate whether CCE training improves emotion regulation and maladaptive mood symptoms.The overarching hypothesis is that training-related improvement in CCE will facilitate improvements in emotion regulation across multiple contexts, and, thus, reduce the symptoms and consequences of emotion dysregulation in bipolar.

The second goal of the project is to collect pilot data, establish feasibility, and gather other information necessary to acquire federal funding for a large-scale, double-blind, randomized control trial of CCE training for bipolar. To ensure subsequent federal funding, the current project design is consistent with an experimental medicine model and NIMH guidelines for clinical trial research. NIMH has a progressive funding structure for the development of novel biological or behavioral interventions. The current project is designed to satisfy requirements of the first phase in this funding structure. Consistent with NIMH guidelines for exploratory clinical trials, the current project has a clearly defined treatment target (i.e. CCE skills) and a theoretical model regarding how the target mechanism is related to psychopathology. The main purpose of an exploratory trial is to verify 'target engagement' - i.e. that the intervention influences the intended treatment target. It is not necessary to have a comparison group. However, evidence of target engagement in a single, active treatment group is a requirement for obtaining more advanced levels of NIMH funding. The current project will evaluate target engagement in a single group that completes CCE training. The study maximize the potential to detect target engagement by using behavioral and neural measures of CCE that are valid, reliable, and sensitive to treatment-related improvement.

Another purpose of the exploratory phase is to gather information about feasibility, tolerability, dose, and other potential factors that could influence treatment effectiveness, patient compliance, and broad implementation, particularly in non-academic settings. Data from the current project will address these issues and provide salient information to guide treatment development and implementation in the next phase. This information includes data on participants' motivation to continue training, enjoyment of training exercises, compliance to the training schedule (e.g. number of days missed, real or perceived obstacles to training, strategies that enhance motivation and compliance, etc.).

In summary, the investigators will conduct an exploratory clinical trial that is consistent with NIMH guidelines for clinical trial research and addresses the goals of an initial (first phase) NIMH grant for novel interventions. Results from the study will provide the pilot data necessary to obtain additional funding for the next phase of treatment development - i.e. An "Exploratory/Developmental Grant for Novel Interventions Phase II (R33)" or a "Confirmatory Efficacy Clinical Trial of Non-Pharmacological Interventions for Mental Disorders (R01)".

ELIGIBILITY:
Inclusion/Exclusion Criteria for All Participants Inclusion Criteria.

At the time of the consent, the subject MUST:

1. be between 18 and 30 years old, inclusive.
2. have learned English before the age of 12.
3. demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in this research study.

Exclusion Criteria.

At the time of the consent, the subject should NOT:

1. have a history of mental retardation (determined by an IQ<70 based on the WRAT or an equivalent brief IQ test) or pervasive developmental disorder; or other neurological disorder (e.g., epilepsy, Parkinson's disease), or another major medical illness.
2. have a current or recent (within past three months) substance use disorder that is characterized as severe as defined by the DSM-5 criteria and confirmed by the SCID-I or by a score of 37 or more on the AADIS.
3. have had, according to the Traumatic Brain Injury (TBI) interview, a moderate or severe TBI where consciousness is lost for 30 minutes or more, or had three or more mild TBIs where consciousness was lost for more than five minutes on each occasion.
4. have severe and persistent ADHD that was diagnosed in childhood (before the age of 12). Subjects who received a diagnosis of ADHD with onset concurrent with bipolar disorder and/or after age 12, will NOT be excluded.
5. have answered 'yes' to Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the C-SSRS or have answered 'yes' to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the C-SSRS "Suicidal Behavior" portion shall be excluded from the study if ideation or behavior occurred within two months of consent. Subjects excluded for this reason will be referred for appropriate treatment.

Additionally, subjects who appear to be intoxicated or under the influence of a controlled substance on any day of assessment must be rescheduled or discontinued based upon the discretion of the staff evaluator.

Additional Inclusion/Exclusion Criteria Specific to Bipolar I Participants Inclusion Criteria. At the time of the consent, the subject MUST

1. meet criteria for Bipolar I Disorder, that is not better explained by another psychiatric disorder, including but not limited to a psychotic disorder, substance-induced bipolar disorder, and bipolar disorder due to a medical condition as defined by DSM5 criteria and confirmed by the SCID.
2. have an onset of Bipolar I Disorder within the past five (5) years, with onset being determined by the first time the subject met DSM-5 criteria for Bipolar I Disorder in their lifetime, as determined by the SCID and regardless of a formal diagnosis.
3. receive a score of less than eight (8) on the YMRS and a score of less than 15 on the MADRS according to the Bipolar Inventory of Symptoms Scale (BISS) at the consent visit.
4. have the visual, auditory, and motor capacity to use the computerized intervention in the judgment of the consenting study staff person.

Exclusion Criteria.

At the time of the consent, the subject should NOT:

1. be in an active illness phase that requires monitoring, intervention, and/or increased psychiatric oversight. Increased psychiatric oversight, may include, but is not limited to:

   1. having had a psychiatric hospitalization in the eight (8) weeks prior to consent.
   2. changes in psychiatric medication in the eight (8) weeks prior to consent.
   3. experiencing four (4) or more episodes of mania and/or depression within the 12 months (i.e. rapid cycling) prior to consent.
2. meet DSM-5 criteria for an episode of mania, hypomania, or depression in the eight (8) weeks prior to consent.
3. have a medication regime consisting of more than four (4) psychotropic medications OR with a high anticholinergic load, defined as benzotropine equivalent greater than two (2) milligrams (Minzenburg et al 2004).
4. have a history of electric convulsive therapy (ECT), transcranial magnetic stimulation (TMS), or deep brain stimulation (DBS).
5. have been treated within 5 years of the date of consent with a computer-based cognitive training program
6. be participating in a concurrent clinical trial that, in the judgment of the staff evaluator could affect the outcome of this one.

Additional Inclusion/Exclusion Criteria Specific to Healthy Subjects Inclusion Criteria.

At the time of the consent, the subject MUST:

1. have no evidence of past history of manic and/or hypomanic episodes as determined by the clinician and described by DSM Criterion A for each type of episode

1. Manic Episode, Criterion A: A distinct period of abnormally and persistently elevated, expansive, or irritable mood and abnormally and persistently increased activity or energy, lasting at least 1 week and present most of the day, nearly every day (or any duration if hospitalization is necessary).
2. Hypomanic Episode, Criterion A: A distinct period of abnormally and persistently elevated, expansive, or irritable mood and abnormally and persistently increased activity or energy, lasting at least 4 consecutive days and present most of the day, nearly every day.

Exclusion Criteria

At the time of the consent, the subject should NOT:

1. meet for a DSM psychiatric disorder, in the last three months
2. have met for a major depressive episode (MDE) in the last year and/or three or more MDEs in their lifetime
3. be receiving current behavioral treatment focusing on emotion regulation or mood problems (e.g. anger management) and/or psychopharmacological treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of CCE training program | 4 weeks
  Participants completed the Intrinsic Motivation Questionnaire to assess enjoyment, usability, and motivation. Rating scale is 1 to 7. An average rating of 4 or above is taken as evidence of feasibility.
Change in Cognitive Control of Emotion (CCE) | 4 weeks
  A main outcome measure for the study is the Change (from pre-to-post intervention) in Cognitive Control of Emotion (CCE) skills. CCE skills are assessed using the appropriate performance metric for each CCE training exercise (e.g. reaction time, accuracy, number of objects remembered, etc.). Individual performance on each of the 5 CCE exercises is measured at the first session of the intervention (i.e. baseline performance) and after the 20th session (approx 4 weeks). Change in CCE is calculated by subtracting the individual's pre-intervention/baseline score from their post-intervention score (i.e. Post intervention score - Pre intervention score = Change Score). One-sample t-tests are used to determine whether the Change Score is significantly different than zero. A significant result indicates that the intervention program had an effect on CCE - the targeted cognitive process.

CONTACTS AND LOCATIONS:
Overall Officials: Christine I Hooker, PhD, Principal Investigator — Rush University Medical Center; Kristen M Haut, PhD, Study Director — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman EG, Hedeker D, Peterson JL, Davis JM. The Altman Self-Rating Mania Scale. Biol Psychiatry. 1997 Nov 15;42(10):948-55. doi: 10.1016/S0006-3223(96)00548-3. PMID 9359982
- [Background] Arbuthnott K, Frank J. Trail making test, part B as a measure of executive control: validation using a set-switching paradigm. J Clin Exp Neuropsychol. 2000 Aug;22(4):518-28. doi: 10.1076/1380-3395(200008)22:4;1-0;FT518. PMID 10923061
- [Background] Bowden CL, Singh V, Thompson P, Gonzalez JM, Katz MM, Dahl M, Prihoda TJ, Chang X. Development of the bipolar inventory of symptoms scale. Acta Psychiatr Scand. 2007 Sep;116(3):189-94. doi: 10.1111/j.1600-0447.2006.00955.x. PMID 17655560
- [Background] Burdick KE, Ketter TA, Goldberg JF, Calabrese JR. Assessing cognitive function in bipolar disorder: challenges and recommendations for clinical trial design. J Clin Psychiatry. 2015 Mar;76(3):e342-50. doi: 10.4088/JCP.14cs09399. PMID 25830456
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carver CS, Ganellen RJ. Depression and components of self-punitiveness: high standards, self-criticism, and overgeneralization. J Abnorm Psychol. 1983 Aug;92(3):330-7. doi: 10.1037//0021-843x.92.3.330. No abstract available. PMID 6619408
- [Background] Carver CS, Johnson SL. Tendencies Toward Mania and Tendencies Toward Depression Have Distinct Motivational, Affective, and Cognitive Correlates. Cognit Ther Res. 2009 Dec;33(6):552-569. doi: 10.1007/s10608-008-9213-y. PMID 20376291
- [Background] Carver, C.S., White, T.L., 1994. Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: the BIS/BAS scales. J. Pers. Soc. Psychol. 67, 319-333.
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629